CLINICAL TRIAL: NCT02376881
Title: Erythropoietin in Methanol Associated Optic Neuropathy
Brief Title: Erythropoietin in Methanol Associated Optic Neuropathy: A Phase-2 Clinical Trial (EPO-MAON Study)
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tehran University of Medical Sciences (Other)
Collaborators: Iran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Farzad Pakdel, Prof., Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ERS139
Record Dates: First submitted 2015-02-17; First posted 2015-03-03 (Estimated); Last update posted 2020-03-10 (Actual); Status verified 2020-03

CONDITIONS: Optic Nerve Diseases
Keywords: Erythropoietin -Methanol - Optic Neuropathy
MeSH Terms: conditions — Optic Nerve Diseases | interventions — Erythropoietin

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- EPO (Experimental): 20,000 IU recombinant human erythropoietin IV infusion in 100 ml normal saline in 2 hr for 3 successive days
  Interventions: Drug: Erythropoietin
- control group (Placebo Comparator): 100 ml normal saline in 2 hr for 3 successive days
  Interventions: Other: placebo

INTERVENTIONS:
Drug: Erythropoietin — 20,000 IU epo IV infusion in 100 ml normal saline in 2 hr for 3 successive days
  Arms: EPO
Other: placebo — 100 ml normal saline in 2 hr for 3 successive days
  Arms: control group

SUMMARY:
Methanol poisoning could result in severe optic neuropathy, profound visual loss and finally optic atrophy and permanent, irreversible optic atrophy and visual loss. Erythropoietin (EPO) has recently emerged as a drug that may help retinal ganglion cell loss and improve optic nerve function in some acquired types of optic neuropathy including traumatic optic neuropathy ,ischemic optic neuropathy and optic neuritis .It has been found that EPO offer some protection to the optic nerve and retina when they are injured and apoptosis process starts in retinal ganglion cells. The standard treatments of methanol poisoning are reanimation, metabolic stabilization, and inhibition of alcohol dehydrogenase by antagonist agents and elimination of toxic metabolites in early phase of toxicity by dialysis. However, after established optic neuropathy and visual loss there is little chance, if any, for visual recovery and no definitive treatment exist for treatment in these cases. The investigators recently reported the investigators preliminary results on 16 cases with methanol poisoning and found a beneficial effect of systemic erythropoietin in methanol associated optic neuropathy. Now, the investigators aim to investigate the effect of this agent in a clinical trial.

The purpose of this study is to determine if EPO could improves optic nerve function and help patients to improve visual recovery after methanol poisoning. Primary outcome measure would be best-corrected visual function and secondary outcome measure is ocular coherence tomography (OCT) measure of mean peripapillary nerve fiber layer thickness. Results of this study could be very valuable in formulating an evidence-based management of Methanol Associated Optic Neuropathy(MAON) and provide a high level evidence for changing the practice on management of methanol poisoning . Also it could provide valuable data for neuroprotective effects of erythropoietin specifically in neuroscience and ophthalmology.

The EPO-MAON trial is designed as a randomized, controlled, observer, and interpreter blinded mono-center pilot trial with two parallel groups and a primary endpoint of best corrected visual acuity during 120 days after enrollment into treatment groups.

All patients with methanol poisoning referred to Farabi hospital will be examined and evaluated for best-corrected visual acuity, pupillary light reflexes, relative afferent pupillary defect, color vision (Ishihara plates), fundus photography, slit lamp exam of anterior segment and fundus exam with 78 D lens.

ELIGIBILITY:
Inclusion Criteria:

1. Patients with confirmed MAON
2. age 10-50 years old
3. Best Corrected Visual Acuity(BCVA)<20/30 or Visual field defect in 10 degrees of central fixation shown in visual field perimetry C-24 SITA(Swedish interactive threshold algorithm)
4. those who can respond to questions and undergo diagnostic tests.

Exclusion Criteria:

1. previous intra-ocular or ocular surface surgeries;
2. those who do not agree to perform ophthalmic exams explained to them by the examiner ophthalmologists
3. those who have history of diabetes mellitus, cardiovascular disease, cerebrovascular disease.
4. Those who had received corticosteroid within past 1 month.
5. Those who has any cornea, lens, retina, optic nerve, choroid or central nervous system(CNS) disease that could potentially affect visual function.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24 (Estimated)
Dates: Start 2015-03; Primary Completion 2019-03-30 (Actual); Study Completion 2020-03-30 (Estimated)

PRIMARY OUTCOMES:
Best Corrected Visual Acuity | changes from baseline at week 12
  centra visual acuity changes from baseline by C Landolt chart after refractive error correction and pinhole if not corrected by glasses alone-converted to logMAR by special prepared table

SECONDARY OUTCOMES:
peripapillary nerve fiber layer thickness | changes from baseline at week 12
  thickness of peripapillary nerve fiber layer using spectral domain OCT

CONTACTS AND LOCATIONS:
Locations (1):
- Farabi Hospital, Tehran University of Medical Sciences, Tehran, Iran

IPD SHARING:
Plan to Share IPD: Undecided